CLINICAL TRIAL: NCT01096576
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of the Dengue Virus Polymerase Inhibitor (Balapiravir) in Male Patients With Confirmed Dengue Virus Infection
Brief Title: A Study of Balapiravir in Patients With Dengue Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PP22799
Record Dates: First submitted 2010-03-17; First posted 2010-03-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Dengue
MeSH Terms: conditions — Dengue | interventions — balapiravir

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: balapiravir [RO4588161]
- B (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: balapiravir [RO4588161] — sequential cohorts receiving doses orally twice daily for 5 days
  Arms: A
Drug: placebo — orally twice daily for 5 days
  Arms: B

SUMMARY:
This randomized, double-blind, multiple-dose, placebo-controlled study will evaluate the safety, tolerability and efficacy of balapiravir in adult male patients with confirmed dengue virus infection whose symptoms began within the 48 hours preceding the first administration of balapiravir. Patients will be randomized to receive either balapiravir or placebo, orally twice daily for 5 days. Anticipated time on treatment as in-patient is 7 days, with an out-patient follow-up to week 12. Target sample size is <200

ELIGIBILITY:
Inclusion Criteria:

* male patients, 18-65 years of age
* dengue virus infection (confirmed by NS1 strip test) with symptom onset </=48 hours before first study drug administration
* patients and their partners of childbearing potential must use 2 forms of contraception until 3 months after receiving the last dose of study drug
* BMI between 18 and 35

Exclusion Criteria:

* positive test at screening for HIV using point of care test, or known HIV infection
* history of any disease known to cause significant alteration in immunologic function or autoimmune disease
* patients taking steroid or other immuno-suppressive therapies
* positive test for drugs of abuse or alcohol using point of care test
* clinically significant abnormal laboratory test results which are deemed unassociated with dengue infection or, alternatively, are diagnostic of dengue shock syndrome

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-07; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability: Adverse events, laboratory parameters, vital signs | days 1-7 and on follow-up days 14, 28 and 84

SECONDARY OUTCOMES:
Viral load | days 1-7 and 14
Pharmacokinetics: plasma concentrations of RO1042897, balapiravir and metabolites | multiple sampling days 1 and 5
Body temperature | days 1-7 and on follow-up days 14, 28 and 84
Immunological parameters: plasma samples (cytokines) | days 1-7 and 14
Hematological parameters: blood samples (red and white blood cell count, hemoglobin, hematocrit, reticulocyte count, fibrinogen, platelet count) | days 1-7, and on follow-up days 14, 28 and 84
Quality of life | assessments days 1, 3, 5, 7, 14, 28 and 84

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Nguyen NM, Tran CN, Phung LK, Duong KT, Huynh Hle A, Farrar J, Nguyen QT, Tran HT, Nguyen CV, Merson L, Hoang LT, Hibberd ML, Aw PP, Wilm A, Nagarajan N, Nguyen DT, Pham MP, Nguyen TT, Javanbakht H, Klumpp K, Hammond J, Petric R, Wolbers M, Nguyen CT, Simmons CP. A randomized, double-blind placebo controlled trial of balapiravir, a polymerase inhibitor, in adult dengue patients. J Infect Dis. 2013 May 1;207(9):1442-50. doi: 10.1093/infdis/jis470. Epub 2012 Jul 17. PMID 22807519